CLINICAL TRIAL: NCT02082756
Title: Effects of Berberine Hydrochloride and Bifidobacterium in Prediabetes Prevention and Treatment：an Open-label, Multicenter，Randomized, Prospective，Controlled Study
Brief Title: Effects of Berberine Hydrochloride and Bifidobacterium in Prediabetes Prevention and Treatment
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: The sponsor have not enough money to support this trial
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2013KTZB03-02-01B
Record Dates: First submitted 2014-03-06; First posted 2014-03-10 (Estimated); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Prediabetes
Keywords: Prediabetes; Berberine Hydrochloride; Bifidobacterium
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Bifidobacterium viable pharmaceutics (Experimental): Bifidobacterium viable pharmaceutics, 2 Capsules, 2/day, 12 weeks
  Interventions: Drug: Bifidobacterium viable pharmaceutics
- Berberine Hydrochloride (Experimental): Berberine Hydrochloride, 0.5g, 2/day, 12 weeks
  Interventions: Drug: Berberine Hydrochloride
- lifestyle counseling (No Intervention)

INTERVENTIONS:
Drug: Bifidobacterium viable pharmaceutics
  Arms: Bifidobacterium viable pharmaceutics
Drug: Berberine Hydrochloride
  Arms: Berberine Hydrochloride

SUMMARY:
The aim of this study is to assess the beneficial effects of Bifidobacterium and Berberine Hydrochloride on lowering glucose and delaying progress to diabetes in patients with prediabetes and to detect the potential mechanism.

DETAILED DESCRIPTION:
Gut microbiota may play an important role in patients with prediabetes. Berberine, which is usually used as an antibiotic drug, has been reported a potential glucose-lowering effect in vitro and in vivo studies. Bifidobacterium, as a familiar probiotics, can modulate gut microbiota and improve glucose and lipid metabolism in animal experiments. Therefore, the aim of this study is to assess the beneficial effects of Bifidobacterium and Berberine Hydrochloride on lowering glucose and delaying progress to diabetes in patients with prediabetes and to detect the potential mechanism.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any trial-related activities
* Male or female between 18 and 70 years of age
* 19≤Body mass index(BMI)≤30kg/m2
* No participate in any clinical trial at least 3 months
* Fasting blood glucose(FBG)<7.0mmol/L and 2-hour postprandial blood glucose(2hPBG)<11.1mmol/L
* Females in child-bearing period should be given birth control
* No severe disease about heart, lung and kidney
* Ability and willingness to adhere to the protocol including performance of self-monitored blood glucose (SMBG) profiles according to the protocol;
* Subject is likely to comply with the Investigators instruction.

Exclusion Criteria:

* Type 2 diabetes mellitus or type 1 diabetes mellitus
* Females of childbearing potential who are pregnant，breastfeeding or intend to become pregnant or are not using adequate contraceptive methods
* Impaired liver function, defined as Aspartate aminotransferase(AST) or Alanine transaminase(ALT)> 2 times upper limit of normal (central laboratory)
* Impaired renal function, defined as serum-creatinine≥133μmol/L
* Uncontrolled treated/untreated severe hypertension (systolic blood pressure≥160mmHg and /or diastolic blood pressure≥95mmHg)
* Chronic gastrointestinal diseases
* Cancer and medical history of cancer (except basal cell skin cancer or squamous cell skin cancer)
* Any clinically significant disease or disorder, which in the Investigator's opinion could interfere with the results of the trial
* Mental incapacity, psychiatric disorder, unwillingness or language barriers precluding adequate understanding or co-operation, including subjects not able to read and write
* Previous participation in this trial. Participation is defined as randomized. Re-screening of screening failures is allowed only once within the limits of the recruitment period
* Known or suspected hypersensitivity to trial products or related products
* Known or suspected abuse of alcohol, narcotics or illicit drugs.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-11 (Estimated); Primary Completion 2018-04 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Change in 2-hour postprandial blood glucose between baseline to week 12 | Baseline and Week 12
  2-hour postprandial blood glucose are measured at baseline and week 12 during a 2 hour-meal test.

SECONDARY OUTCOMES:
Gut microbiome composition | Baseline and week 12
  Faecal bacterial composition determined from microbiological cultures and deep metagenomic next-generation sequencing of bacterial DNA in feces.
Adverse effects | From baseline to week 12
  Standardized questionaries regarding gastrointestinal function are filled out at each study visit (0, 4, 8 and 12 weeks after randomization) to detect possible adverse effects of antibiotics. In addition, subjects are given a calendar and informed to write down any symptom or illness during the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Qiu Ji, Ph.D..M.D., Principal Investigator — Department of Endocrinology, Xijing Hospital, Fourth Military Medical University
Locations (4):
- China (4):
  - Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - The 323rd Hospital of People's Liberation Army, Xi'an, Shaanxi
  - First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Shaanxi Provincial People's Hospital, Xi'an, Shaanxi